CLINICAL TRIAL: NCT01602445
Title: Analysis of Pro-coagulant and Thrombin-generation Markers for the Prediction of Therapeutic Failure in Cancer Patients at Risk for Recurrence of Venous Thromboembolism: A Pilot Study
Brief Title: Pro-coagulant Markers and Anticoagulant Failure in Cancer Patients at Risk for Recurrence of Venous Thromboembolism
Acronym: REMARK
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: HSFO-000524; 20120208-01H (Other: Ottawa Hospital Research Ethics Board)
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Venous Thromboembolism; Deep-Vein Thrombosis; Pulmonary Embolism; Cancer
Keywords: Venous Thrombosis; Coagulation factors; Cancer; Blood
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum specimens Optional DNA banking
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients: All cancer patients with a diagnosed acute symptomatic VTE episode.

SUMMARY:
The presence of clots in the veins of arms and/or legs or lungs of Cancer patients decreases their quality of life, delays their treatment and may cause death. The best way to avoid new clots is by giving blood thinners before clots are formed, but even some patients who are taking blood thinners may form blood clots. A major problem is that it is difficult to know which patients form clots while they are receiving blood thinners, a situation called treatment failure. Several studies have shown that by doing blood tests that measure the formation of clots, the investigators could know if the patient is responding to the blood thinners. If this is proven, the investigators will be able to apply these tests to all patients.

DETAILED DESCRIPTION:
Therapeutic failure in cancer patients at high risk for recurrence of Venous thromboembolism (VTE) may be as high as 20% and the risk of death from a recurrent episode of pulmonary embolism is at least 8%. Studies that have used pro-coagulant and thrombin generation markers support the notion that cancer is associated with a hypercoagulability state and that intensified doses of anticoagulation may be necessary to suppress this state. Thus, it may be possible that by using these tests, we would identify the patients that do not respond to standard doses of anticoagulation. To date, only few small studies have evaluated the use of pro-coagulant markers in cancer patients but this data is promising. Our study will measure pro-coagulant markers in cancer patients at risk for VTE recurrence to determine if there is a relationship between the changes in the levels of pro-coagulant markers and VTE recurrence while taking anticoagulation with low-molecular weight-heparin (LMWH). The evaluation of the pro-coagulant markers may enable new treatment strategies in cancer patients who fail their initial treatment. Patients will be stratified by a risk model developed by our group and will be validate with this study. This new approach has the potential to improve the recovery of patients, to reduce death and disability due to clots in the veins of legs or arms and/or lungs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any type of cancer (except basal cell and squamous cell carcinoma of the skin) and at any stage of the disease or treatment
* Confirmed newly diagnosed acute symptomatic VTE (proximal DVT, PE, Arm DVT, Multiple SSPE only)
* Planned treatment of VTE with low-molecular weight heparin (LMWH)
* Age 18 years old or older.

Exclusion Criteria:

* Planned cell transplant
* Patient receiving anticoagulation due to other clinical indications
* Patient who has received more than one therapeutic dose of LMWH
* Unable or unwilling to provide written, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referrals of cancer patients to the Thrombosis clinic at each participating center at the time that an acute episode of VTE has been confirmed ( within 0 +/- 1 day) from the start of anticoagulation treatment. Our centers provide VTE treatment for all the cancer patients in our regions given the design of the Ontario Cancer Program, ensuring a generalizable patient population.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Relative changes on biochemical markers | at initiation of anticoagulation (baseline); at 7-14 days; 21-35 days; 37- 44 days; 83-97 days; and 173-187 days after initiation of anticoagulation.
  The following pro-coagulant and thrombin-generation markers will be measured:
  1. Prothrombin fragments F1+2;
  2. D-dimer,
  3. thrombin-antithrombin (TAT)
  4. Soluble P-selectin.
  For each patient, we will calculate baseline values and the relative changes (delta) of procoagulant and thrombin generation markers. The relative changes (delta) will be defined by the percentage of change in the marker at each visit relative to baseline measurement.

SECONDARY OUTCOMES:
Rates of treatment failure | 6 months
  This outcome will be measured by the proportion of cancer patients who might develop recurrent VTE while on 6-month treatment with anticoagulation within the time-frame of the study.
Correlation between treatment failure and markers | 6 months after treatment failure
  This outcome will be assessed by determining the best cutoff for each marker that would correctly classify success or failure to anticoagulation treatment
Compliance to anticoagulation treatment | 6 months
  Compliance to medication will be measured by review of the patient medication diary.

CONTACTS AND LOCATIONS:
Overall Officials: Philip S Wells, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - Capital Health District Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Science Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - CHUM-Notre-Dame Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noble S, Pasi J. Epidemiology and pathophysiology of cancer-associated thrombosis. Br J Cancer. 2010 Apr 13;102 Suppl 1(Suppl 1):S2-9. doi: 10.1038/sj.bjc.6605599. PMID 20386546
- [Background] Blom JW, Vanderschoot JP, Oostindier MJ, Osanto S, van der Meer FJ, Rosendaal FR. Incidence of venous thrombosis in a large cohort of 66,329 cancer patients: results of a record linkage study. J Thromb Haemost. 2006 Mar;4(3):529-35. doi: 10.1111/j.1538-7836.2006.01804.x. PMID 16460435
- [Background] Prandoni P, Lensing AW, Piccioli A, Bernardi E, Simioni P, Girolami B, Marchiori A, Sabbion P, Prins MH, Noventa F, Girolami A. Recurrent venous thromboembolism and bleeding complications during anticoagulant treatment in patients with cancer and venous thrombosis. Blood. 2002 Nov 15;100(10):3484-8. doi: 10.1182/blood-2002-01-0108. Epub 2002 Jul 12. PMID 12393647
- [Background] Coleman R, MacCallum P. Treatment and secondary prevention of venous thromboembolism in cancer. Br J Cancer. 2010 Apr 13;102 Suppl 1(Suppl 1):S17-23. doi: 10.1038/sj.bjc.6605601. PMID 20386545
- [Background] Lee AY, Levine MN, Baker RI, Bowden C, Kakkar AK, Prins M, Rickles FR, Julian JA, Haley S, Kovacs MJ, Gent M; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low-molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med. 2003 Jul 10;349(2):146-53. doi: 10.1056/NEJMoa025313. PMID 12853587
- [Background] Weitz IC, Israel VK, Waisman JR, Presant CA, Rochanda L, Liebman HA. Chemotherapy-induced activation of hemostasis: effect of a low molecular weight heparin (dalteparin sodium) on plasma markers of hemostatic activation. Thromb Haemost. 2002 Aug;88(2):213-20. PMID 12195692
- [Background] Traby L, Kaider A, Schmid R, Kranz A, Quehenberger P, Kyrle PA, Eichinger S. The effects of low-molecular-weight heparin at two different dosages on thrombin generation in cancer patients. A randomised controlled trial. Thromb Haemost. 2010 Jul;104(1):92-9. doi: 10.1160/TH09-12-0863. Epub 2010 May 10. PMID 20458441
- [Background] Kirwan CC, McDowell G, McCollum CN, Kumar S, Byrne GJ. Early changes in the haemostatic and procoagulant systems after chemotherapy for breast cancer. Br J Cancer. 2008 Oct 7;99(7):1000-6. doi: 10.1038/sj.bjc.6604620. Epub 2008 Sep 2. PMID 18766191
- [Result] Louzada ML, Carrier M, Lazo-Langner A, Dao V, Zhang J, Kovacs MJ, Lee AY, Levine MN, Meyer G, Rodger M, Wells PS. Validation of a clinical prediction rule for risk stratification of recurrent venous thromboembolism in patients with cancer-associated venous thromboembolism. American Society of Hematology, 52nd Annual Meeting, Orlando Florida, December 4-7, 2010. Abstract 4209. Poster Board III-988.
- [Result] Louzada ML, Carrier M, Lazo-Langner A, Dao V, Kovacs MJ, Ramsay TO, Rodger MA, Zhang J, Lee AY, Meyer G, Wells PS. Development of a clinical prediction rule for risk stratification of recurrent venous thromboembolism in patients with cancer-associated venous thromboembolism. Circulation. 2012 Jul 24;126(4):448-54. doi: 10.1161/CIRCULATIONAHA.111.051920. Epub 2012 Jun 7. PMID 22679142